CLINICAL TRIAL: NCT04469751
Title: Correlation Between Dorsalis Pedis and Radial Arterial Invasive Blood Pressures During Anesthesia Induction in Neurosurgical Patients A Self-control Study
Brief Title: Correlation Between Dorsalis Pedis and Radial Arterial Invasive Blood Pressures During Anesthesia Induction in Neurosurgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-511
Record Dates: First submitted 2020-07-05; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Blood Pressure
Keywords: correlation radial artery dorsalis pedis artery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients undergoing neurosurgery (Experimental): radial artery and dorsalis pedis artery intubated with BD Insyte-W 22G artery puncture needle under local anaesthesia
  Interventions: Diagnostic Test: invasive blood pressure monitoring

INTERVENTIONS:
Diagnostic Test: invasive blood pressure monitoring — radial artery and dorsalis pedis artery intubated with BD Insyte-W 22G artery puncture needle under local anaesthesia

SUMMARY:
Anesthesiologists need to understand the specific difference between dorsalis pedis arterial(DPA) pressure and the more commonly used radial arterial(RA) pressure When blood pressure monitoring at DPA. Generally, the systolic blood pressure measured in DPA is significantly higher than that in RA, with little difference of diastolic blood pressure and mean artery pressure in two sites. However, there is no specific study on the difference between them, and it is not clear how the diagnosis and treatment threshold should be adjusted when relying on DPA blood pressure measurement to guide treatment. The intraoperative blood pressure of patients is in the normal range in most cases. The purpose of this study is to analyze the correlation of different blood pressure stratification (RASBP90-109mmHg,110-129mmHg,130-149mmHg) of DPA-RA in the normal range to understand the correlation of DPA-RA in different blood pressure ranges, to provide a reference for clinical decision-making and hemodynamic management.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent neurosurgery,American Society of Anesthesiologists' physical status 1-3, BMI 18-24 kg/m², a clinical need for invasive arterial pressure monitoring in the supine position.

Exclusion Criteria:

* Arterial puncture site injury or infection,heart failure, severe arrhythmia, congenital heart disease, hypertension, diabetes,preoperative use of dehydration, and intracranial hypertension drugs such as mannitol, peripheral and macrovascular diseases, chronic lung disease, history of heart or lung surgery, The Allens test was positive.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
DPA-RA invasive blood pressure | During anesthesia induction
  All DPA-RA blood pressure dates are Separate analyzed in the following three intervals: Group1 (RASBP 90-109mmHg), Group1 (RASBP 110-129mmHg), Group1 (RASBP 130-149mmHg).The correlation and consistency of each group were analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

REFERENCES:
- [Background] Chen Y, Cui J, Sun JJ, Wang E, Zhu Y, Li Y, Lu K. Gradient between dorsalis pedis and radial arterial blood pressures during sevoflurane anaesthesia: A self-control study in patients undergoing neurosurgery. Eur J Anaesthesiol. 2016 Feb;33(2):110-7. doi: 10.1097/EJA.0000000000000295. PMID 26694940
- [Background] Chen Y, Wang E, Zhu Y, Li Y, Lu K. Dorsalis pedis arterial pressure is lower than noninvasive arm blood pressure in normotensive patients under sevoflurane anesthesia. Blood Press Monit. 2016 Feb;21(1):27-32. doi: 10.1097/MBP.0000000000000153. PMID 26484744